CLINICAL TRIAL: NCT04860687
Title: Quality of Life After COVID-19 Related Acute respIratory Distress Syndrome Among ICU Survivors Patients in Italy: the ODISSEA Study.
Acronym: ODISSEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: ODISSEA 1.0
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Post Traumatic Stress Disorder; Quality of Life
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory insufficiency is one of the principal causes of intensive care admission for COVID 19 positive patients. This may determine a variable mortality rate ranging from 25-30%.

In these patients, many days of non-invasive or invasive mechanical ventilation are needed to correct severe hypoxemia.

Mechanical ventilation is not a direct therapy but allows the clinicians to prolong the "time-to-recovery" interval necessary for COVID 19 respiratory insufficiency treatment.

Long intensive care stay, mechanical ventilation, the use of steroids and sedatives have an impact on the survivors.

Previous studies demonstrated that patients admitted to intensive care with non-COVID acute respiratory distress syndrome had a reduction in the quality of life even up to one year after discharge.

The aim of this study is to understand if COVID-19 related acute respiratory distress syndrome has a worse impact on the quality of life one year after discharge when compared with non-COVID-19 acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients discharged from the intensive care unit after admission for COVID-19 respiratory insufficiency that requested non-invasive or invasive mechanical ventilation

Exclusion Criteria:

* history of dementia
* history of behavior disorders
* pre-existing tracheostomy
* advanced oncologic disease
* end-stage-organ disease (dialysis, or enlisted for organ transplantation)
* no consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID 19 positive patients admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 309 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey 36 | One year after discharge
  Evaluate the physical abilities of patients discharged from the intensive care unit after admission for COVID-19 respiratory insufficiency. The scale ranges from 0 to 100, where 0 is the worse value and 100 is the best.

SECONDARY OUTCOMES:
Impact of Event Scale - Revised (IES-R) | One year after discharge
  Identify post traumatic stress disorder in patients discharged from the intensive care unit after admission for COVID-19 respiratory insufficiency. The scale ranges from 0 to 88, where 0 is the best value and 88 the worst.
Age | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the age of the patients
Gender | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the gender of the patients
Scholarship | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the scholarship of the patients
Marital status | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the marital status of the patients
Steroids | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the use of steroids
Muscle relaxants | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the use of muscle relaxants
Renal replacement therapy | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with the use of renal replacement therapy
Tracheostomy | One year after discharge
  Evaluate if there is an association between quality of life measured with Short Form Health Survey 36 scale and Impact of Event Scale - Revised and post traumatic stress disorder with tracheostomy

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Anesthesia and Intensive Care, Academic Hospital of Catanzaro, Catanzaro, Calabria
  - Anesthesia, Intensive Care and Pain Therapy, Academic Hospital "Federico II" of Naples, Naples, Campania
  - Anesthesia and Intensive Care, Academic Hospital of Ferrara, Ferrara, Emilia-Romagna
  - Anesthesia and Intensive Care 2, Academic Hospital of Parma, Parma, Emilia-Romagna
  - Anesthesia and Intensive Care Department, Ravenna Hospital, Ravenna, Emilia-Romagna
  - Department of Anesthesia and Intensive Care, Academic Hospital of Udine, Udine, Friuli Venezia Giulia
  - Anesthesia and Intensive Care 1, Hospital of Trento, Trento, Trentino-Alto Adige
  - Anesthesia and Intensive Care 2, Perugia Hospital, Perugia, Umbria

REFERENCES:
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Azoulay E, Thiery G, Chevret S, Moreau D, Darmon M, Bergeron A, Yang K, Meignin V, Ciroldi M, Le Gall JR, Tazi A, Schlemmer B. The prognosis of acute respiratory failure in critically ill cancer patients. Medicine (Baltimore). 2004 Nov;83(6):360-370. doi: 10.1097/01.md.0000145370.63676.fb. PMID 15525848
- [Background] Thiery G, Azoulay E, Darmon M, Ciroldi M, De Miranda S, Levy V, Fieux F, Moreau D, Le Gall JR, Schlemmer B. Outcome of cancer patients considered for intensive care unit admission: a hospital-wide prospective study. J Clin Oncol. 2005 Jul 1;23(19):4406-13. doi: 10.1200/JCO.2005.01.487. PMID 15994150
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Vetrugno L, Bove T, Orso D, Barbariol F, Bassi F, Boero E, Ferrari G, Kong R. Our Italian experience using lung ultrasound for identification, grading and serial follow-up of severity of lung involvement for management of patients with COVID-19. Echocardiography. 2020 Apr;37(4):625-627. doi: 10.1111/echo.14664. Epub 2020 Apr 15. PMID 32239532
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Derived] Vetrugno L, Sala A, Deana C, Meroi F, Grandesso M, Maggiore SM, Isola M, De Martino M, Restaino S, Vizzielli G, Bove T, Driul L. Quality of life 1 year after hospital discharge in unvaccinated pregnant women with COVID-19 respiratory symptoms: a prospective observational study (ODISSEA-PINK study). Front Med (Lausanne). 2023 Sep 6;10:1225648. doi: 10.3389/fmed.2023.1225648. eCollection 2023. PMID 37746068